CLINICAL TRIAL: NCT02320188
Title: Effect of Eccentric Exercise Training in Rheumatoid Cachexia
Brief Title: Eccentric Exercise and Cachexia in Rheumatoid Arthritis
Acronym: EECRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0215; 2013-A01789-36 (Other: CHU de Clermont-Ferrand)
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis
Keywords: modification of treatment planned; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

ARMS (3):
- Eccentric exercise (Experimental): Thirty sessions of Eccentric training in twelve weeks. Average of two sessions per week without spacing higher than eight days between two sessions.
  Interventions: Other: Eccentric exercise
- Concentric exercise (Experimental): Thirty sessions of Concentric training in twelve weeks. Average of three sessions per week without spacing higher than eight days between two sessions.
  Interventions: Other: Concentric exercise
- No training (control) (No Intervention): Usual activities. No further training during the observation period

INTERVENTIONS:
Other: Eccentric exercise — This study aimed to determine the muscle effects of ECC training, with the primary outcome being the knee extensor strength gain at 3 months.
  Arms: Eccentric exercise
Other: Concentric exercise — The purpose of the study is to determine in a randomized controlled trial (RCT), the efficacy of eccentric exercise training in restoring muscle mass and function in patients with rheumatoid cachexia.
  Arms: Concentric exercise

SUMMARY:
The purpose of the study is to determine in a randomized controlled trial (RCT), the efficacy of eccentric exercise training in restoring muscle mass and function in patients with rheumatoid cachexia.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is characterized by severe disability and metabolic changes leading to an increase in cardiovascular mortality compared with the general population. RA is an independent cardiovascular risk factor. In contrast to the general population, RA patients with low body mass index (BMI) had a significantly higher risk of cardiovascular death. Low BMI may indicate rheumatoid cachexia and may explain the excess cardiovascular risk and mortality. Cachexia is defined by is a loss of body cell mass, predominantly in skeletal muscle, associated with increased fat mass and often stable weight. Rheumatoid cachexia, not well recognized, is frequent, affecting two third of patients. Pathogenesis may include inflammatory cytokine production, physical inactivity, higher catabolism and reduced peripheral insulin action. Therapeutic strategy includes increasing physical activity and the treatment of disease itself. Studies have shown that regular progressive resistance strength training improves strength and pain in patients with well-controlled RA without exacerbating disease activity or joint pain. At comparable mechanical power output, eccentric (ECC ) exercises are characterised by lower metabolic demand than concentric (CON) exercises. ECC exercise is characterised not only by its low energy cost, but also by specific cardiocirculatory specificity. In patients with Parkinson's disease, compared to a conventional rehabilitation programme, ECC training better improved quadriceps muscle volume. In overweight and diabetic patients, ECC training improved resting energy expenditure and fat oxidation, blood lipid profile and insulin resistance compared to CON training. As in cancers, ECC training appears to be particularly suitable for patients with rheumatoid cachexia as it can maximize the functional and structural muscle responses with low energy cost populations.

This study aimed to determine the muscle effects of ECC training, with the primary outcome being the knee extensor strength gain at 3 months. Secondary outcomes are the improvement in muscle mass, functional status and cardiovascular risk. From patients who consented in ECC training group, muscle biopsy specimens from vastus lateralis will be obtained at baseline prior to the training period. Primary and secondary outcome criteria will be assessed at inclusion, at 3 months, and 6 months.

In total, 48 patients will need to be recruited. These patients will be randomly assigned to one of the 3 groups, with each group comprising 16 patients: group 1 with ECC training, group 2 with CONC training, group 3 with no training (control). The training program will consist in 30 sessions over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 66 years old
* Diagnosis of rheumatoid arthritis according to ACR 1987 or ACR/EULAR 2010 criteria
* Activity of the disease measured by the DAS28 ≤3.2
* Stable for at least 3 months, no modification of treatment planned in the 3 months
* Steroids prednisone ≤ 0.1 mg/kg/day
* Steinbrocker functional classification for functional disability ≤ II
* The Questionnaire of Baecke for measurement of physical activity < 7.5
* Stable nutritional diet
* Patients resident in the area of "Grand Clermont"
* Clinical cachexia as defined by upper arm muscle area ≤75th percentile for age and sex

Exclusion Criteria:

* contraindication to exercise or to exercise stress test
* advanced hip or knee osteoarthritis
* Planned surgery of hip or knee
* Hip or knee arthroplasty preventing pedaling
* Chronic disease associated with cachexia
* Nutritional intervention
* Pregnancy
* For muscle biopsy: contraindication to local anesthesia, anticoagulation therapy

Ages: 40 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Isometric knee extensor strength gain measured by an isokinetic dynamometer | at 3 months

SECONDARY OUTCOMES:
improvement in muscle mass | Up to 30 days before the beginning of the training, after 3 and 6 months
  quadriceps muscle volume
improvement in fonctional status | At the beginning of the training, after 3 and 6 months
  Body composition : Lean body mass, Appendicular lean mass
improvement in cardiovascular risk | At the beginning of the training, after 3 and 6 months
  Cardiovascular risk : arterial compliance

CONTACTS AND LOCATIONS:
Overall Officials: Anne TOURNADRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France